CLINICAL TRIAL: NCT03736811
Title: Nonabsorbable Versus Absorbable Sutures for Anterior Colporrhaphy: a Randomized Controlled Trial
Brief Title: Nonabsorbable Versus Absorbable Sutures for Anterior Colporrhaphy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Myung Jae Jeon, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNUH-1810-037-977
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Absorbable suture (Active Comparator): will undergo anterior colporrhaphy in a traditional manner using either 2-0 polyglactin 910 [Vicryl] or polydioxanone [PDS II] sutures.
  Interventions: Device: Polyglactin 910 or polydioxanone
- Nonabsorbable suture (Experimental): will undergo anterior colporrhaphy in a traditional manner using either 2-0 polyester [Ethibond Excel] or polypropylene [Prolene] sutures.
  Interventions: Device: Polyester or polypropylene

INTERVENTIONS:
Device: Polyglactin 910 or polydioxanone — Vicryl or PDS II
  Arms: Absorbable suture
Device: Polyester or polypropylene — Ethibond Excel or prolene
  Arms: Nonabsorbable suture

SUMMARY:
The objective of this is to compare surgical outcomes of anterior colporrhaphy using nonabsorbable sutures with anterior colporrhaphy using absorbable sutures.

DETAILED DESCRIPTION:
This trial is a prospective, randomized trial conducted with the aim to determine superiority of anterior colporrhaphy using nonabsorbable sutures over absorbable sutures with regard to the primary outcome. Participants will undergo reconstructive surgery for prolapse, including anterior colporrhaphy using the assigned suture materials under general or spinal anesthesia. The anterior colporrhaphy will be performed in a traditional manner with midline plication of the fibromuscular layer using either 2-0 nonabsorbable (polyester or polypropylene; Ethicon, Somerville, NJ) or absorbable (polyglactin 910 or polydioxanone; Ethicon) sutures. Concomitant procedures will be performed as intended prior to surgery. Women with a uterus in situ will undergo hysterectomy and all women will receive an apical suspension procedure, including uterosacral ligament suspension, sacrospinous ligament fixation, and iliococcygeal suspension, according to the preference of surgeon. Posterior colporrhaphy and incontinence surgery will also be performed, if indicated (i.e. women with Bp ≥-1 or documented urodynamic stress incontinence).

Enrollment, treatment and data collection will be standardized by all sites. The study will be a single-blind study, as it is impossible to blind the study surgeon for the surgical procedure to which the subject in assigned. However, all outcomes assessors and the subjects will be blinded to the treatment assignment. Postoperative follow-up will take place after 5 weeks, 6 months and 12 months. Patients will undergo a standard gynecological examination including POPQ and fill in questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Anterior vaginal descent beyond the hymen (i.e. POPQ Ba>0)
* Vaginal bulge symptoms (i.e. an affirmative response to the question 3 from the PFDI-20)
* Reconstructive surgery is planned

Exclusion Criteria:

* Recurrent anterior vaginal wall prolapse
* Reconstructive surgery using mesh or obliterative surgery for prolapse is planned
* Known pelvic malignancy
* Systemic glucocorticoid or immunosuppressant treatment
* Subject wishes to retain her uterus
* Subject is unable and unwilling to participate in

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Surgical success | One year after surgery
  defined as the absence of all of the following: (1) anterior vaginal descent beyond the hymen (POPQ point Ba>0); (2) presence of vaginal bulge symptoms (affirmative response to the question 3 from the Pelvic Floor Distress Inventory-20 ("do you usually have a bulge or something falling out that you can see or feel in your vaginal area?"; (3) re-treatment for recurrent anterior vaginal wall prolapse by either surgery or pessary.

SECONDARY OUTCOMES:
The rate of anterior vaginal descent beyond the hymen | One year after surgery
  POPQ point Ba>0
The rate of vaginal bulge symptoms | One year after surgery
  an affirmative response to the question 3 from PFDI-20
The rate of re-treatment for recurrent anterior vaginal wall prolapse | One year after surgery
  by either surgery or pessary
The rate of suboptimal anatomical outcome in each compartment | One year after surgery
  POPQ point Ba, C, or Bp ≥-1
Change of POPQ values | From baseline to 1 year after surgery
  point Ba, C, Bp and TVL
Change of PFDI-20 scores | From baseline to 1 year after surgery
  The PFDI-20 is a valid and reliable condition-specific quality-of-life questionnaires for women with pelvic floor disorders. It has 20 items and 3 scales (Pelvic Organ Prolapse Distress Inventory, Colorectal-Anal Distress Inventory and Urinary Distress Inventory). Each scale is scored from 0 to 100; higher scores indicate greater symptom burden.
  The PFDI-20 total score is obtained by adding the scores from the 3 scale scores together (0-300).
The rate of adverse events related with anterior colporrhaphy | From baseline to 1 year after surgery
  1. intraoperative- bladder injury, ureteral obstruction, massive bleeding
  2. postoperative- hematoma, vesico-vaginal fistula, ureteral obstruction, urinary tract infection, incomplete bladder emptying, overactive bladder or stress incontinence symptoms, suture erosion, vaginal wound dehiscence, infection or granulation tissue, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Myung Jae Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Myung Jae, Jeon, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeon MJ, Suh DH, Kim CH, Cho HH, Shin JH, Lee SR, Jung YW, Kim SR, Kong MK. Non-absorbable versus absorbable sutures for anterior colporrhaphy: study protocol for a randomised controlled trial in South Korea. BMJ Open. 2020 Jun 16;10(6):e034218. doi: 10.1136/bmjopen-2019-034218. PMID 32554735